CLINICAL TRIAL: NCT00003742
Title: Phase I Trial of Paclitaxel, Cisplatin, and Irinotecan in Patients With Advanced Solid Tumor Malignancies
Brief Title: Combination Chemotherapy in Treating Patients With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 98-100; CDR0000066860 (Registry Identifier: PDQ (Physician Data Query)); NCI-G99-1495
Record Dates: First submitted 1999-11-01; First posted 2004-03-15 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Cisplatin; Irinotecan; Paclitaxel

INTERVENTIONS:
Drug: cisplatin
Drug: irinotecan hydrochloride
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combination chemotherapy in treating patients with locally advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of paclitaxel when combined with cisplatin and irinotecan in patients with locally advanced or metastatic solid tumors. II. Determine the dose limiting toxicity of paclitaxel when combined with cisplatin and irinotecan in this patient population. III. Establish the recommended phase II dose for this regimen in this patient population. IV. Assess the antitumor activity of this regimen in selected solid tumor malignancies.

OUTLINE: This is a dose escalation study of paclitaxel. All patients receive paclitaxel IV over 1 hour, then cisplatin IV over 30 minutes, followed by irinotecan IV over 30 minutes weekly for 4 weeks on days 1, 8, 15, and 22. Treatment is repeated every six weeks for at least 3 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of paclitaxel. If 2 or more patients experience dose limiting toxicity (DLT) at a particular dose level, escalation ceases and the maximum tolerated dose (MTD) is defined as the previous dose level. Patients are followed until death.

PROJECTED ACCRUAL: Approximately 12-27 patients will be accrued for this study within 6-9 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven locally advanced (unresectable or recurrent) or metastatic solid tumor No bone metastases, abnormal radionuclide bone scan or pleural effusions as the sole indicators of disease No CNS metastases or carcinomatous meningitis

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL AST no greater than 3 times upper limit of normal (ULN) (no greater than 5 times ULN if liver metastases present) No Gilbert's Disease Renal: Creatinine no greater than 1.5 mg/dL Serum calcium less than 12.0 mg/dL No symptomatic hypercalcemia Cardiovascular: No unstable angina No active angina No New York Heart Association class III or IV heart disease No uncontrolled asymptomatic congestive cardiac failure At least 6 months since any myocardial infarction Pulmonary: No interstitial pulmonary fibrosis Other: No history of seizure disorder and receiving phenytoin, phenobarbital, or other antiepileptic medication No active or uncontrolled infection No uncontrolled diabetes mellitus Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: One prior chemotherapy regimen allowed Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy and recovered No prior mantle, hemibody, pelvic, or lumbar spine irradiation Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-10; Primary Completion 2001-08 (Actual); Study Completion 2001-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H. Ilson, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States